CLINICAL TRIAL: NCT04566406
Title: Risk Factors for Hemodynamic Instability During Laparoscopic Pheochromocytoma Resection - Single Centre Experience
Brief Title: Pheochromocytoma and Hemodynamic Instability
Status: Completed | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Karolina Zawadzka, Principal Investigator, Jagiellonian University
Other Study IDs: Pheochromocytoma&HI
Record Dates: First submitted 2020-09-17; First posted 2020-09-28 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Pheochromocytoma; Hypertension; Surgery
Keywords: pheochromocytoma; laparoscopy; haemodynamics; surgery
MeSH Terms: conditions — Pheochromocytoma; Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Laparoscopic adrenalectomy — Preoperative staging in all cases consisted of computed tomography or/and magnetic resonance imaging. Prior to surgery, a routine panel of laboratory tests was carried out. The catecholamines metabolites (metanephrine, normetanephrine, and methoxytyramine) were measured from 24-hour urine collection. All patients were preoperatively treated with phenoxybenzamine or alternative doxazosin.Additionally, beta-blockers in case of coexisting tachycardia were given. In the morning of the operation, preinduction blood pressure was measured. Pneumoperitoneum was achieved by insufflating CO2 gas to an intraperitoneal pressure of 12 mmHg. The operative method in our department was laparoscopic transperitoneal lateral total adrenalectomy. Intraoperatively SBP and diastolic blood pressure (DBP) were measured and recorded every 10 minutes. To treat hypertensive and hypotensive episodes, intravenous doses of urapidil, ephedrine, nitrates, MgSO4, norepinephrine, or ß-blockers were administered.

SUMMARY:
The aims of our study were to define perioperative HI during laparoscopic adrenalectomy for pheochromocytoma, assess the incidence of perioperative HI, and identify predictive factors of perioperative HI in our group of patients.

DETAILED DESCRIPTION:
The study was a retrospective observation of consecutive patients with histologically confirmed pheochromocytoma undergoing laparoscopic adrenalectomy between years 2003 and 2019.

ELIGIBILITY:
Inclusion Criteria:

* patients with histologically confirmed pheochromocytoma undergoing laparoscopic adrenalectomy

Exclusion Criteria:

* bilateral tumour
* no histopathological result
* neoplastic spread

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with histologically confirmed pheochromocytoma undergoing laparoscopic adrenalectomy
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2003-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Hemodynamic Instability (n, %) | intraoperative
  Hemodynamic instability was defined as an occurrence of both intraoperative episodes of systolic blood pressure above 160 mm Hg and vasoactive (vasodilators or vasoconstrictors) drugs administration. Patients were divided into two groups: one which met both above criteria, and another one without hemodynamic instability.

SECONDARY OUTCOMES:
Number of Complications in Patients (n, %) | Within 30 days after surgery
  Data on morbidity were classified according to the Clavien-Dindo classification.
Number of Cardiovascular Complications in Patients (n, %) | Within 30 days after surgery
  Cardiovascular morbidity was defined as postoperative morbidity related to the cardiovascular system: postoperative hypotensive or hypertensive episodes requiring pharmacologic treatment, need for blood transfusion, myocardial or digestive ischemia, stroke, and postoperative hospitalization in intensive care unit (ICU) for cardiac-related causes.

OTHER OUTCOMES:
Length of hospital stay (days) | Up to 30 days
Duration of anaesthesia (min) | Intraoperative
Duration of surgery (min) | Intraoperative
Patients needing blood transfusion, n (%) | Intraoperative
Mean intraoperative blood loss (ml) | Intraoperative
Number of participants who required intraoperative vasodilators administration (n, %) | Intraoperative
Number of participants who required intraoperative vasopressors administration (n, %) | Intraoperative
Patients with episodes systolic blood pressure >200 mmHg (n, %) | Intraoperative
Patients with episodes systolic blood pressure >180 mmHg (n, %) | Intraoperative
Patients with episodes systolic blood pressure >160 mmHg (n, %) | Intraoperative
Number of participants who required postoperative vasopressorss administration (n, %) | Within 24 hours after surgery

IPD SHARING:
Plan to Share IPD: No